CLINICAL TRIAL: NCT03140540
Title: Transesophageal Echocardiography as a Guide for Fluid Optimization in Major Abdominal Oncosurgery
Brief Title: TEE as a Guide for Fluid Optimization in Major Abdominal Oncosurgery
Acronym: VTI SVV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr soumi pathak, Principal Investigator, Rajiv Gandhi Cancer Institute & Research Center, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RGCI ID:500/AN/ANK-02
Record Dates: First submitted 2017-04-15; First posted 2017-05-04 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Fluid Therapy
Keywords: Fluid management; goal-directed therapy; transesophageal echocardiography

STUDY DESIGN:
Intervention Model Description: TEE as guide for tailoring perioperative fluid therapy to achieve individualized hemodynamic endpoint , target hemodynamic goals of stroke volume index (SVI) greater than 35 mL/m2 and cardiac index greater than 2.5 L/min/m2 and tissue oxygen delivery. Lactate levels as a surrogate indicator of organ perfusion as measured by arterial blood gas analysis intraoperatively , after 12 hours and 48 hrs postoperatively.
Who Masked: Care Provider
Masking Description: The intensivist taking care of the patient postoperatively not aware of the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (stroke volume variation) guided fluid (Active Comparator): Stroke volume variation guided intraoperative intravenous fluid will be administered.
  Interventions: Other: Stroke volume variation guided intravenous fluid.
- Group B(Study group) TEE guided fluid (Active Comparator): Transesophageal echocardiography will be used to guide the fluid therapy.
  Interventions: Other: TEE guided fluid therapy will be administered

INTERVENTIONS:
Other: TEE guided fluid therapy will be administered — Transesophageal echocardiography will be used to guide the fluid therapy. Velocity time integral of aorta <20 ,200ml colloid bolus to be administered.
  Arms: Group B(Study group) TEE guided fluid
Other: Stroke volume variation guided intravenous fluid. — Active Comparator: Group A control group (SVV guided fluid ) Stroke volume variation guided intraoperative intravenous fluid will be administered. SVV >10, 200 ml of colloid bolus to be given
  Arms: Group A (stroke volume variation) guided fluid

SUMMARY:
Transesophageal echocardiography (TEE) as guide for tailoring perioperative fluid therapy to achieve individualized hemodynamic endpoint, target hemodynamic goals of stroke volume index (SVI) greater than 35 mL/m2 and cardiac index greater than 2.5 L/min/m2 and tissue oxygen delivery.

Lactate levels as a surrogate indicator of organ perfusion as measured by arterial blood gas analysis intraoperatively, after 12 hours and 48 hrs postoperatively

DETAILED DESCRIPTION:
TEE as guide for tailoring perioperative fluid therapy to achieve target hemodynamic goals of stroke volume index (SVI) greater than 35 mL/m2 and cardiac index greater than 2.5 L/min/m2 and tissue oxygen delivery.

GDT (goal directed therapy): continuous infusion of crystalloids 2 mL/kg/h.

If (velocity time integral) VTI <20, 250 mL colloid bolus administered. Dose repeated every 10 min until goal of VTI >20 met. Norepinephrine titrated to maintain MAP(mean arterial pressure) > 65 mm Hg. Blood transfused for haemoglobin <8 g Lactate levels as a surrogate indicator of organ perfusion as measured by arterial blood gas analysis at time of incision intraoperatively and after 12 hours and 48 hrs. The incidence of postoperative complications, morbidity, mortality, duration of mechanical ventilation and ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1, 2 and 3
* Undergoing major abdominal oncosurgery

Exclusion Criteria:

* Any contraindication for TEE probe insertion as oesophageal varices , oesophageal and gastric carcinoma , severe left ventricular hypertrophy , coagulopathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-16 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 48 hours
  The incidence of postoperative complications in percentage

SECONDARY OUTCOMES:
intraoperative fluid | intraoperative period (hours)
  Amount of intraoperative fluid in litres to be compared
median icu stay | 1 week
  duration of icu stay

CONTACTS AND LOCATIONS:
Locations (1):
- Rajiv Gandhi Cancer Institute, Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guarracino F. [The role of transesophageal echocardiography in intraoperative hemodynamic monitoring]. Minerva Anestesiol. 2001 Apr;67(4):320-4. Italian. PMID 11376533
- [Result] Trinooson CD, Gold ME. Impact of goal-directed perioperative fluid management in high-risk surgical procedures: a literature review. AANA J. 2013 Oct;81(5):357-68. PMID 24354071